CLINICAL TRIAL: NCT03354949
Title: Postural Wheelchair Control in Hemiplegic Stroke Patients
Brief Title: Base Positioning Wheelchair Hemiplegic
Status: Completed | Type: Observational
Sponsor: Groupement Hospitalier Intercommunal du Vexin (Other)
Responsible Party: Sponsor
Other Study IDs: GHIV0117
Record Dates: First submitted 2017-11-17; First posted 2017-11-28 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Wheelchair
Keywords: Wheelchair; Hemiplegia; Stroke; Postural control; Pain
MeSH Terms: conditions — Hemiplegia; Stroke; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Positioning hemiplegic.: Positioning all hemiplegic by stroke requiring a single wheelchair even at the exit of the SSR and hemiplegic patient with sequelae.
  Measurement of sitting postural control of the adult (MCPAA). Assessment of wheelchair pain in the spine and ischia by a self-evaluation scale (EVA).
  Propulsion speed of a wheelchair.
  Interventions: Other: Measurement of sitting postural control of the adult (MCPAA)

INTERVENTIONS:
Other: Measurement of sitting postural control of the adult (MCPAA) — The Adult Seated Postural Control Measure 2.0 (MCPAA 2.0) is a clinical evaluation tool for sitting postural control of adult clients using a locomotion aid. It thus allows the evaluation of the two variables inherent to the postural control sit, the alignment of body segments and the influence between movement and posture.
  It can also be used to evaluate the changes in seated postural control due to changes over time or to an adaptation of the sitting posture.
  Assessment of wheelchair pain in the spine and ischia by a self-evaluation scale (EVA).
  the speed of propulsion by a wheelchair.

SUMMARY:
The investigators looked at the population of hemiplegic stroke participants hospitalized with GHIV : the investigators assessed the postural control of the participants of the chair using MCPAA, and assessed the pain of the participants while sitting in a wheelchair. The investigators then had to the participants try positioning equipment and then prescribed it once the choice was made. The investigators then reassessed postural control and wheelchair pain with this positioning equipment.

DETAILED DESCRIPTION:
For each hemiplegic participants with wheelchair user stroke, the investigators collect : date of birth, date of stroke, side of hemiplegia. The wheelchair propulsion mode, the degree of autonomy (FAC and Enjalber scales), the way bed - wheelchair transfers are made. Assessment of wheelchair pain in the spine and Ischia with EVA. Time to travel 10 meters in a wheelchair. Postural control of the wheelchair is evaluated by the MCPAA. The investigators then carry out tests of positioning equipment : backrest, cushion, form elements and belt. This material is tried for several days. If it is appropriate (improvement on the postural control and on the pains), otherwise another material is tried.

When the choice is made, the material is prescribed. The participant is seen again 3 months after the delivery of his personal material, and the same evaluation is redone.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegia by stroke
* Wheelchair user

Exclusion Criteria:

* Two-handed propulsion of the wheelchair
* Cognitive impairment preventing clinical examination

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Positioning of all hemiplegics by stroke requiring a wheelchair even punctual at the exit of the SSR compared to patients with hemiplegic sequelae.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Study the improvement of the basin retroversion. | Through study completion, an average of one year.
  The Adult Seated Postural Control Measure 2.0 (MCPAA 2.0) is a clinical evaluation tool for sitting postural control of adult clients using a locomotion aid. It thus allows the evaluation of the two variables inherent to the postural control sit, the alignment of body segments and the influence between movement and posture. It can also be used to evaluate the changes in seated postural control due to changes over time or to an adaptation of the sitting posture.

SECONDARY OUTCOMES:
The tilt. | Through study completion, an average of one year.
  Assessment of wheelchair pain in the spine and ischia by a self-evaluation scale (EVA). The self-evaluation scale (EVA) is used to assess participant pain.
  It is in the form of a straight line of 100 mm. This scale is composed on the reverse side of a horizontal line from "no pain" to "maximum pain imaginable". The left side corresponds to "no pain", the right end corresponds to "maximum pain imaginable". The participant indicates, with the cursor, his level of pain on the line. The pain score is displayed on the front of the scale.
Propulsion speed. | Through study completion, an average of one year.
  The propelling speed of the wheelchair.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine PELLIGRINI, Principal Investigator — Groupe Hospitalier Intercommunal du Vexin

IPD SHARING:
Plan to Share IPD: No